CLINICAL TRIAL: NCT07230795
Title: AI-informed Colorectal Cancer (CRC) Screening Navigation vs. Standard of Care Among Screening-naive Penn Medicine Patients 45-49 Years Old to Increase CRC Screening Uptake
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09225; 858875 (Other: Penn IRB)
Record Dates: First submitted 2025-09-08; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Navigator Assistance (Experimental): A trained CRC navigator who will conduct outreach and navigation by interviewing these patients according to a script that consists of a statement of research, confirms eligibility, communicates their relative increased risk of CRC, assesses and addresses barriers to completion of CRC screening, and offers an adapted validated questionnaire regarding these barriers for patients to complete asynchronously. The navigator will be able to address barriers such as lack of awareness/knowledge about screening, misinformation, negative attitudes and fear, scheduling, inability to afford the prep, and lack of transportation and escort. The calls performed by the patient navigator will not be recorded.
  Interventions: Other: Intervention Arm
- Control Arm - NO Navigator Assistance (No Intervention): Patients in the control arm will be enrolled under a waiver. They will only receive standard of care.

INTERVENTIONS:
Other: Intervention Arm — The intervention arm will consist of a trained CRC navigator who will conduct outreach and navigation by interviewing these patients according to a script that consists of a statement of research, confirms eligibility, communicates their relative increased risk of CRC, assesses and addresses barriers to completion of CRC screening, and offers an adapted validated questionnaire regarding these barriers for patients to complete asynchronously. The navigator will be able to address barriers such as lack of awareness/knowledge about screening, misinformation, negative attitudes and fear, scheduling, inability to afford the prep, and lack of transportation and escort. The calls performed by the patient navigator will not be recorded.
  Other Names: Patient navigator
  Arms: Intervention Arm - Navigator Assistance

SUMMARY:
This project aims to use machine learning algorithms (MLA) to identify and risk-stratify individuals between the ages of 45-49 who are more likely to have colorectal pathology and merit prioritized CRC screening and patient navigation. Patients deemed to be at higher risk for CRC by MLA will be randomized to an intervention group to receive risk-informed patient navigation and a usual care control group. The patient navigation will assist in completing either a fecal immunochemical test (FIT) or a colonoscopy. For the usual care control group, patients may still receive patient navigation for colonoscopy assistance. A referral to a nurse navigator can be initiated by a healthcare staff member in the following ways: 1) procedure scheduling staff will provide navigator's contact number if the patient expresses difficulty with obtaining a ride home 2) endoscopy staff and physicians can message navigator electronically 3) PCPs can place a navigation order in the EHR for patients deemed to need additional support such as with prep, education, transportation 4) providers will directly contact the director of the navigation system (Dr. Carmen Guerra) for referral.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-49
2. Not up to date with CRC screening within the recommended period of time (colonoscopy within 10 years, FIT within 1 year, Cologuard within 3 years, sigmoidoscopy within 3-5 years)
3. Have primary care providers in Penn Internal Medicine and Family Medicine Practices
4. Have at least 1 outpatient CBC in the past 12 months.

Exclusion Criteria:

1. Prior history of CRC
2. Late-stage cancer of any organ (stage 4)
3. History of colectomy
4. Demonstrated high-risk of colorectal cancer (e.g. inflammatory bowel disease, hereditary colorectal cancer syndromes)

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7120 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment in the Navigator program | 12 month
  The patient navigation will assist in completing their colorectal cancer screening. The only test are either a fecal immunochemical test (FIT) or a colonoscopy. No other tests are required.
Completion of colonoscopy or FIT testing | 12 month
  The patient navigation will assist in completing either a fecal immunochemical test (FIT) or a colonoscopy. The only test are either a fecal immunochemical test (FIT) or a colonoscopy. No other tests are required.
Abnormal screening findings (positive FIT, abnormal colonoscopy findings). S | 12 month
  We will evaluate the effectiveness of the program on uptake of navigation and completion of CRC screening, rates of abnormal screening results, abnormal stool test follow-up with diagnostic colonoscopy, time to screening uptake, and CRC and precancerous lesion detection.

SECONDARY OUTCOMES:
Screening uptake | Firtst 3 month
  We will evaluate the effectiveness of the program on the uptake of navigation.
Colonoscopy follow-up for abnormal FIT | Firtst 3 month
  We will evaluate the effectiveness of the program on the uptake of navigation and completion of colorectal cancer screening.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No